CLINICAL TRIAL: NCT06787625
Title: Pilot Feasibility Study for the Development of Organoids From Primary Colorectal Tumors and Synchronous Liver Metastases
Brief Title: Development of Organoids From Primary Colorectal Tumors and Synchronous Liver Metastases
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS87/IRE/24
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Colo-rectal Cancer
Keywords: colororectal cancer; organoids
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — colorectal tumor tissue samples, liver metastases tissue samples, whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pilot feasibility study for the development of organoids from primary colorectal tumors and synchronous liver metastases, to prepare organoids from primary colorectal tumors and synchronous liver metastases. The organoids will allow us to study the function of genes targeted by the activity of the NF-Y/p53 complex.

DETAILED DESCRIPTION:
Organoids will allow us to study the function of genes that are targets of the NF-Y/p53 complex activity. In these organoids, we will perform overexpression and/or silencing of these genes and assays of proliferation, invasion and motility. We will also perform functional assays in cocultures of the organoids with PBMCs from the same patients. This could allow the discovery of new pathways that could be targeted by targeted therapy and/or immunotherapy. Organoid preparation will be performed from fresh colorectal cancer tissue and liver metastasis following enzymatic digestion. Organoid culture medium and specific organic matrix will be used

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Histological and cytological diagnosis of colorectal cancer neoplasia that has developed a liver metastasis
* Patients who are candidates for surgery for colorectal cancer with liver metastasis
* Signing of the relevant informed consent form.

Exclusion Criteria:

* All exclusion criteria adopted in surgical protocols will be applied to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancer and synchronous liver metastases who will undergo liver resection surgery
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-05-25 (Actual); Primary Completion 2028-01-25 (Estimated); Study Completion 2028-05-25 (Estimated)

PRIMARY OUTCOMES:
Descriptive analyses | 36 months
  Given the pilot nature of the study, we will only perform descriptive analyses, overexpression or silencing experiments of target genes of the NF-Y/p53 complex activity. These experiments will indicate the impact on the viability of the organoid of target genes of the NF-Y/p53 complex activity. All the variables of interest will be summarized through absolute frequencies and percentages, if categorical or through medians and relative range, if continuous.

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Piaggio, Biologist, Principal Investigator — IRCCS National Cancer Institute
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy